CLINICAL TRIAL: NCT06023823
Title: Dry Needling of the Abductor Hallucis Muscle in the Management of Hallux Valgus; Effect on Pain, Function and Valgus Angle
Brief Title: The Role of Dry Needling in Hallux Valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Tayyip Dede, Medical Doctor, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07/04/2023; 2011-KAEK-50;88
Record Dates: First submitted 2023-08-26; First posted 2023-09-05 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Hallux Valgus; Myofascial Pain Syndrome
MeSH Terms: conditions — Hallux Valgus; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toe spread out treatment (Active Comparator)
  Interventions: Other: Toe spread out; Other: Dry needling+Toe spread out
- Dry needling (Active Comparator)
  Interventions: Other: Dry needling+Toe spread out

INTERVENTIONS:
Other: Toe spread out — toe-spread-out exercise.
  Arms: Toe spread out treatment
Other: Dry needling+Toe spread out — The group will be given 3 sessions of dry needling with Seirin branded 0.6*50 mm acupuncture needles for trigger pointe in the abductor hallucis muscle and additionally toe-spread-out exercise.

SUMMARY:
Forty Hallux valgus patients between the ages of 25-65 years, who are admitted to the Physical Medicine and Rehabilitation clinic with the complaint of 1st Metatarsophalangeal (MTF) pain and who meet the inclusion and exclusion criteria will be included. Hallux valgus (HV) angles will be measured by dorsoplantar radiography before the patients start the study. The HV angle was measured as the angle between the bisection line of the first metatarsal bone and the first proximal phalanx. Demographic data (age, gender, body mass index) will be recorded at the beginning of the study. Then, the initial Foot Functional Index (FFI) and Visual Analog Scale (VAS) scales were completed. The 1st MTF joint angle was also measured with a goniometer and recorded before starting the study. The patients were divided into two groups. The first group will be given 3 sessions of dry needling with Seirin branded 0.6*50 mm acupuncture needles for trigger point in the abductor hallucis muscle and toe-spread-out exercise. The second group will receive only toe-spread-out exercises. After starting the treatment, FFI and VAS scores and 1st MTF angles will be measured and recorded weekly with a goniometer. At the end of the 3-week treatment, the FFI and VAS scores of the participants will be re-evaluated after 1 week and 1 month, and the participants will be re-evaluated with a goniometer. The hallux valgus angle will be re-evaluated with X-ray 4 weeks after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 25-65 years old with pain for more than 4 weeks
* Hallux valgus angle between 16-40 degrees
* Activity VAS value above 4

Exclusion Criteria:

* Patients diagnosed with rheumatologic diseases
* Those diagnosed with Diabetes Mellitus (DM), those with chronic liver and kidney failure
* Those who received anti-inflammatory-analgesic treatment in the last 1 week
* Diagnosed with inflammatory rheumatic disease
* Those with a history of foot surgery
* Those with mid or hindfoot deformity
* Those with 1st MTF joint problems other than hallux valgus
* Those with a history of orthotic use
* Previous history of central or peripheral nerve damage, lower extremity neuropathy
* Those diagnosed with Diabetes Mellitus
* Those with cognitive impairment
* Unassisted mobilization

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Does dry needling make an additional contribution to the spread out exercise in the pain management of hallux valgus? | Baseline, 3 week, 7 week
  Pain assessment was performed with (Visual Analog Scale) VAS score at baseline, 3.w and 8.w.
Does dry needling make an additional contribution to the spread out exercise in the functional management of hallux valgus? | Baseline, 3 week, 7 week
  Function assessment was performed with (Foot Functional INdex) FFI score at baseline, 3.w and 8.w.
Does dry needling provide an additional contribution to the spread out exercise in the hallux valgus angle? | Baseline, 7 week
  The hallux valgus angle will be measured at baseline and 7.w on direct radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Tayyip Dede, Principal Investigator — İstanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Resarch Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes